CLINICAL TRIAL: NCT06259149
Title: A Study of Initiation Timing of VTE Prevention After Colorectal Cancer Surgery: a Single-center, Prospective, Observational Cohort Study
Brief Title: A Study of Initiation Timing of VTE Prevention After Colorectal Cancer Surgery
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IIT-2023-0295
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: blood and Colorectal cancer tissue
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early initiation of drug prophylaxis (within 24 hours after surgery): Patients who underwent surgery received prophylactic administration of low molecular weight heparin (nardraparin calcium injection) at a time point of 24 hours after surgery，this group carries out early initiation of drug prophylaxis (within 24 hours after surgery)
  Interventions: Drug: Nardraparin calcium injection
- Late initiation of drug prophylaxis (24 hours after surgery): Patients who underwent surgery received prophylactic administration of low molecular weight heparin (nardraparin calcium injection) at a time point of 24 hours after surgery，this group carries out late initiation of drug prophylaxis ( 24 hours after surgery)
  Interventions: Drug: Nardraparin calcium injection

INTERVENTIONS:
Drug: Nardraparin calcium injection — The dose of nardraparin calcium injection is 100AxaIU/kg, adjusted according to the patient's body weight, and is injected subcutaneously once a day

SUMMARY:
This project intends to conduct a single-center, prospective, observational cohort study to explore the impact of the timing of drug prophylaxis on the risk of postoperative bleeding and the preventive effect of VTE in the prevention and management of postoperative venous thromboembolism (VTE) after colorectal cancer (CRC) surgery in Chinese population, and to determine its application and promotion value. The research results of this project can provide useful reference for optimizing the prevention and management of VTE after CRC operation.

DETAILED DESCRIPTION:
This study is a single-center, prospective, observational cohort study. The design and implementation of the whole study were carried out according to the CONSORT principle. The study was conducted at the Department of Gastrointestinal Surgery, Renji Hospital, Shanghai Jiao Tong University School of Medicine, and patients were followed up for 28 days.

Postoperative patients with colorectal cancer who met the criteria were included. All patients were initiated with low molecular weight heparin (nardraparin calcium injection) for drug prophylaxis after surgery. In clinical practice, patients who underwent surgery at different times on the same day received prophylactic administration of low molecular weight heparin at 24h after surgery, forming two cohorts of early initiation (within 24 hours after surgery) and late initiation (beyond 24 hours after surgery). According to the previous clinical data survey in the past year, since the number of operating tables and the end time of surgery are relatively fixed every day, the number of people in each group of early start and late start groups is about 300 per group per year according to the end time of surgery, which basically conforms to the ratio of 1:1.

The dose of low molecular weight heparin (Nardrheparin calcium injection) was 100AxaIU/kg, adjusted according to the patient's body weight, and was administered subcutaneously once a day throughout the patient's hospital stay. All patients underwent color Doppler ultrasound of lower limbs before discharge (7-10 days after surgery) and 28 days after surgery, including screening for thrombus in the proximal deep vein (femoral vein, popliteal vein), distal deep vein (posterior tibial vein, peroneal vein and muscular vein) and venous communication branch. Each enrolled patient will be followed up for 28 days, and all patients will be followed up 28 days after surgery. If the patient is unable to return to the hospital at the scheduled follow-up time point, the patient can be reminded by phone to be admitted for follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* ① Age > 18 years old;

  ② The patient was diagnosed with colorectal cancer, and the cTMN stage was cT1-2, N0 or cT3, N0 or any cT, N1-2; (3) The patient was diagnosed with colorectal cancer and was able to receive radical surgery (laparoscopic or open surgery). The expected operation time was >45 minutes, and the expected postoperative survival time was >6 months.

  ④ The patient or guardian agrees to the study plan and signs the informed consent.

Exclusion Criteria:

* ① Renal insufficiency (CrCl<30 mL/min) or hepatic insufficiency (ALT> 3 times the upper limit of normal);

  * The patient was diagnosed with colorectal cancer with a cTMN stage of cT4 and/or local unresectable lesions. Unresectable local recurrent lesions included: (1) extensive lateral pelvic wall invasion, (2) external iliac vascular involvement, (3) tumor invasion into the great sciatic notch, sciatic nerve invasion, and (4) invasion of the second sacrum level and above.

Known allergy to low molecular weight heparin (LWMH), narcotic drugs or radiocontrast agents; The presence of systemic hemorrhagic disease or bleeding tendency, such as active peptic ulcer, uncontrolled hypertension, cerebral thrombosis, cerebral hemorrhage or neurosurgical history within 6 months;

* known brain metastases, endocarditis, or history of heparin-induced thrombocytopenia;

  * VTE occurred within 3 months before surgery;

    * Use heparin or oral anticoagulant therapy within 5 days before surgery; Women who are pregnant or breastfeeding;

      * Any situation in which the investigator determines that the subject is not suitable for anticoagulant therapy.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient was diagnosed with colorectal cancer and underwent radical surgery (laparoscopic or open surgery) with an estimated operation time of >45 minutes. Patients with expected survival >6 months after surgery
Sampling Method: Probability Sample
Enrollment: 914 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
VTE events within 28 days after surgery | 7 and 28 days after surgery
  Patients were followed up for VTE events, including deep vein thrombosis (DVT) and pulmonary thromboembolism (PE), within 28 days after surgery. Diagnosis of DVT: The lower limb is examined based on clinical symptoms (swelling and pain in the lower limb, tenderness in the back of the lower limb and/or in the inner thigh) and/or by color ultrasound or venography. The diagnosis of PE is based on clinical findings (dyspnea and shortness of breath), laboratory tests (plasma D-dimer), and CT pulmonary angiography (CTPA). Vte events were evaluated at 7 and 28 days after surgery. If a patient develops a VTE event, the patient is treated with VTE and assessed for thrombotic progression by ultrasound in both lower limb veins after 2 weeks.

SECONDARY OUTCOMES:
Any bleeding event within 28 days after surgery | 1，7 and 28 days after surgery
  Patients were followed up for any bleeding events within 28 days after surgery, including major and minor bleeding events. According to the International Society of Thrombosis and Hemostasis Standards (ISTH standards). All patients were followed up at 1, 7, and 28 days after surgery through inpatient or outpatient follow-up and bleeding investigation.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Chun Gu, Principal Investigator — Department of Pharmacy, Renji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Department of Gastrointestinal Surgery, Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided